CLINICAL TRIAL: NCT06850792
Title: imprOving Adherence to Pulmonary artErial hyperteNsion Treatment With teLemedicIne and patieNt guidaNce - A Multicenter Pre- and Post-intervention Evaluation Study
Brief Title: imprOving Adherence to Pulmonary artErial hyperteNsion Treatment With teLemedicIne and patieNt guidaNce
Acronym: OPENLINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86868325.7.1001
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH); Pulmonary Arterial Hypertension (PAH); Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH); Medication Adherence; Telemedicine; Patient Education; Remote Monitoring; Digital Health Intervention; Randomized Controlled Trial (RCT); Multicenter Study; COMPERA 2.0; REVEAL Lite; Six-Minute Walk Test (6MWT); Quality of Life; CAMPHOR Questionnaire; Martín-Bayarre-Grau (MBG) Scale; Oral Therapy for PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a multicenter, pre-post interventional study evaluating the impact of telemedicine on medication adherence in patients with pulmonary arterial hypertension (PAH) on stable oral therapy. Participants will receive biweekly teleconsultations over 24 weeks, focused on adherence support, education, and symptom management. The primary outcome is change in adherence measured by the Martín-Bayarre-Grau scale. Secondary outcomes include changes in functional class, 6-minute walk distance, BNP levels, risk stratification (COMPERA 2.0, REVEAL Lite), hospitalizations, mortality, and quality of life assessed by the CAMPHOR questionnaire. The study aims to determine whether a structured remote follow-up can enhance adherence and improve clinical outcomes in PAH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine-Based Intervention to Improve Adherence in PAH Patients on Oral Therapy (Experimental): Participants will receive biweekly teleconsultations over 24 weeks, as part of a structured telemedicine intervention to support medication adherence in patients with pulmonary arterial hypertension (PAH) on stable oral therapy. Each teleconsultation is delivered by a trained healthcare professional and includes adherence assessment, identification of barriers, guidance on side effects, educational reinforcement, and motivational support. The intervention does not change the medical regimen but aims to optimize adherence and clinical outcomes through remote follow-up. Data will be collected at baseline and at 24 weeks to evaluate changes in adherence (Martín-Bayarre-Grau scale), functional class, 6-minute walk distance, BNP levels, risk stratification (COMPERA 2.0, REVEAL Lite), hospitalizations, mortality, and quality of life (CAMPHOR).
  Interventions: Behavioral: Telemedicine-Based Adherence Support

INTERVENTIONS:
Behavioral: Telemedicine-Based Adherence Support — The intervention consists of biweekly teleconsultations for six months, conducted by healthcare professionals, focusing on medication adherence, patient education, side effect management, and remote support for individuals with pulmonary arterial hypertension (PAH). Patients will receive structured guidance on treatment adherence, tailored counseling, and real-time problem-solving strategies. The goal is to improve adherence to oral PAH therapy and enhance clinical outcomes compared to standard care.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a progressive condition with high morbidity, frequent hospitalizations, and risk of right heart failure. Despite advances in treatment, poor adherence remains a major challenge. This randomized controlled study assesses whether remote monitoring can improve treatment adherence, clinical outcomes, and side effect management in PAH patients on oral therapy.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a severe, progressive condition requiring strict adherence to complex treatment regimens to improve outcomes. Despite advances in pharmacological therapy, non-adherence remains a significant challenge, impacting disease progression and increasing healthcare burden.

The OPENLINE study is a randomized, multicenter clinical trial designed to evaluate the impact of a structured telemedicine intervention on treatment adherence in PAH patients receiving stable oral therapy. Participants in the intervention group will receive biweekly teleconsultations for six months, focusing on patient education, adherence monitoring, and side effect management. The control group will follow standard clinical care without additional remote support.

The primary outcome is medication adherence, assessed using the Martín-Bayarre-Grau (MBG) scale. Secondary outcomes include changes in functional class, six-minute walk test distance, brain natriuretic peptide (BNP) levels, risk stratification (COMPERA 2.0 and REVEAL Lite), hospitalizations, mortality, and quality of life measured by the CAMPHOR questionnaire.

This study aims to determine whether a telemedicine-based intervention can enhance medication adherence and improve clinical outcomes in PAH patients, potentially informing future care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years diagnosed with pulmonary arterial hypertension (PAH) (Group 1 of the WHO classification).
* Stable oral PAH therapy (including endothelin receptor antagonists, phosphodiesterase-5 inhibitors, or prostacyclin pathway agents) for at least four weeks prior to enrollment.
* Ability to participate in remote teleconsultations (access to a phone or internet).
* Signed informed consent agreeing to study participation.

Exclusion Criteria:

* Severe cognitive impairment or psychiatric disorders that could affect adherence or study participation.
* Inability to communicate via phone or telemedicine due to technical or personal constraints.
* Concurrent participation in another interventional clinical trial that could interfere with outcomes.
* Life expectancy <6 months due to any condition unrelated to PAH.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence (Martín-Bayarre-Grau Scale - MBG) | 24 weeks (end of study period)
  Adherence to oral pulmonary arterial hypertension (PAH) therapy will be evaluated using the Martín-Bayarre-Grau (MBG) scale, a validated questionnaire assessing adherence behaviors such as medication timing, dose compliance, and integration into daily routines. The scale generates a quantitative score ranging from 0 to 100, with higher values reflecting better adherence. The study will compare MBG scores obtained at baseline and after 24 weeks of biweekly teleconsultations to assess the impact of the telemedicine intervention on treatment adherence in a pre-post design.

SECONDARY OUTCOMES:
Functional Class (WHO/NYHA Classification) | 24 weeks
  Functional class will be assessed using the World Health Organization (WHO)/New York Heart Association (NYHA) classification, which categorizes the severity of symptoms and physical activity limitations in patients with pulmonary arterial hypertension (PAH). The classification ranges from Class I (no symptoms) to Class IV (symptoms at rest). Changes in functional class will be evaluated by comparing baseline and 24-week assessments to determine the impact of the telemedicine intervention on clinical status.
Six-Minute Walk Test (6MWT) Distance | 24 weeks
  Distance walked during the six-minute walk test (6MWT) will be measured to evaluate functional capacity and exercise tolerance in patients with pulmonary arterial hypertension (PAH). The test will be conducted at baseline and after 24 weeks of telemedicine follow-up. Changes in the distance walked (in meters) will be analyzed to assess the impact of the intervention on physical performance.
Brain Natriuretic Peptide (BNP) Levels | 24 weeks
  BNP levels, a biomarker for right ventricular function and PAH severity, will be measured at baseline and at 24 weeks to assess changes in cardiac strain.
Risk Stratification (COMPERA 2.0) | 24 weeks
  PAH risk stratification scores using COMPERA 2.0 will be calculated at baseline and at 24 weeks to assess changes in disease severity.
Hospitalizations and Mortality | 24 weeks
  The number of hospitalizations due to PAH-related complications and all-cause mortality will be recorded throughout the 24-week study
Quality of Life (CAMPHOR Questionnaire) | 24 weeks
  Quality of life will be evaluated using the CAMPHOR questionnaire, a validated tool assessing symptoms, activity limitations, and emotional well-being in PAH patients. Changes in scores from baseline to 24 weeks will be analyzed.
Risk Stratification (REVEAL Lite) | 24 weeks
  PAH risk stratification scores using REVEAL LITE will be calculated at baseline and at 24 weeks to assess changes in disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- InCor - Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No